CLINICAL TRIAL: NCT03994874
Title: Peritoneal Ultrafiltration in Cardio Renal Syndrome to Prevent Heart Failure Exacerbation.
Brief Title: Peritoneal Ultrafiltration in Cardio Renal Syndrome.
Acronym: PURE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CQ012019
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-05

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Carnitine; Xylitol

STUDY DESIGN:
Intervention Model Description: Patients will be assigned randomly to receive either PolyCore PUF (over the top of their prescribed heart failure medications), for 6 months, or to the control arm receiving no PUF therapy.
Who Masked: Outcomes Assessor
Masking Description: A blinded independent review committee, comprised of experienced cardiologist and nephrologists, who are non-participating investigators in this study, will be appointed to confirm the primary end-point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PolyCore PUF (Experimental): PolyCore peritoneal ultrafiltration (PUF) (over the top of patient's prescribed heart failure medications), for 6 months.
  Interventions: Drug: PolyCore (Polydextrin, L-Carnitine, D-xylitol)
- Control (No Intervention): Patients in the control arm (receiving no PUF therapy) will remain on their prescribed heart failure medications.

INTERVENTIONS:
Drug: PolyCore (Polydextrin, L-Carnitine, D-xylitol) — A single nightly exchange, with 2 liters PolyCore solution, lasting 12-14 hours. Patients should remain on their prescribed heart failure medications and the same dosing schedule for the duration of the study unless investigators determine medically necessary to change.
  Other Names: PolyCore peritoneal dialysis solution
  Arms: PolyCore PUF

SUMMARY:
Randomized, controlled, unblinded, adaptive design clinical trial to evaluate the safety and efficacy of PolyCore (Polydextrin, L-Carnitine, D-xylitol) peritoneal ultrafiltration (PUF) in patients with heart failure and reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
The study will include adults HFrEF patients, that despite guidelines directed medical therapy still retain a congestive heart failure (HF) picture. During the study, patients should remain on their prescribed heart failure medications and the same dosing schedule for the duration of the study unless investigators determine medically necessary to change. Patients will be assigned randomly to receive either PolyCore PUF (over the top of their prescribed heart failure medications), for 6 months, or to the control arm receiving stable medical therapy according to international guidelines and comprehensive of loop diuretic (furosemide) dose till to 2.5mg/kg/day, without PUF therapy. The PUF ultrafiltration will be performed with a single nightly exchange, with 2 liters PolyCore solution, lasting 12-14 hours, for 6 months. An independent data safety monitoring board (DSMB) will be convened for this study and will review the results of the trial at regular intervals to protect patients participating in the study. An adaptive interim analysis will be performed when in each group 20 patients have completed 6 months in the study, for analysis of the primary outcome. The purpose of the adaptive interim analysis is to calculate the final study sample size.The DSMB will closely examine the interim primary efficacy results, respecting the confidentiality and integrity of data, to investigate the final sample sizes necessary to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 yrs
* Left ventricular ejection fraction ≤60%
* NYHA Classification of III-IV despite guidelines directed medical therapy
* Right ventricular failure due to after load mismatch, addressed by the presence of tricuspid calve regurgitation (≥ moderate) and by the disproportioned increase of the right atrial pressure (RAP) versus the capillary wedge pressure (CWP) with a ratio ≥0.65, detected with right heart catheterization performed after stable medical therapy according to international guidelines and comprehensive of loop diuretic (equivalent to furosemide oral dose till 2.0 mg/kg/day), coupled with urinary sodium excretion ≤ mEq/L, confirmatory of loop diuretic resistance.
* Cava vein enlargement (inner diameter, detected with focused echocardiography, between 1,5 and 2,5 cm, with respiratory collapse <50% or absent due to intravascular fluid overload)
* Decreased kidney function addressed by the measurement of glomerular filtration rate (GFR) urea clearance + creatinine clearance/2 (>15 ml/min/1,73 m2)
* NT pro-BNP plasma concentration > 1000 pg/ml or BNP plasma concentration > 250 pg/ml
* at least one episode of pulmonary or systemic congestion requiring high-dose intravenous diuretics (or diuretic combinations) in the 6 months befor the study enrollment
* An appropriate PUF technique candidate.
* Signed informed consent

Exclusion Criteria:

* Recipients of heart transplantation
* Presence of a mechanical circulatory support device;
* Hypertrophic obstructive cardiomyopathy;
* Uncontrolled hypertension with systolic blood pressure ≥ 160 mmHg
* Severe valvular stenosis;
* Restrictive cardiomyopathy;
* Acute coronary syndrome ≤ 6 months before;
* Active myocarditis
* Cardiosurgical or Endo-radiological heart procedures ≤ 6 months before
* Cardiac resynchronization therapy (CRT) implantation or upgrading of pacemaker (PM) or implantable cardioverter defibrillator (ICD) to CRT ≤ 6 months before;
* Patient with end-stage renal disease, GFR urea clearance + creatinine clearance/2 (<15 ml/min/1,73 m2 GFR)
* Any major organ transplant (liver, lung, kidney)
* Lung embolism ≤ 6 months before;
* Fibrotic lung disease;
* Liver Cirrhosis;
* Absolute contraindication to peritoneal catheter implantation;
* Logistical and or organizational contra-indication to treatment
* Active malignancy;
* Female patients who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical trial and for three months later
* Female patients of childbearing age who do not use adequate contracteption.
* Unwilling and unable to give informed consent;
* Enrolment in another clinical trial involving medical or device based interventions.
* Hypersensibility to IMP components.
* Evidence of any condition that, according to the investigators' judgment, could expose the subject to undue risk and/or prevent the subject from participating in the study procedures and/or potentially afftecting the study quality data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Composite end-point of mortality and worsening patient's condition | Up to 7 months from randomization
  * patient's mortality - or
  * the need of increasing of ≥50% the initial daily dose of loop diuretic - or
  * the hospitalization for infusional therapy with loop diuretic based on the lack of adequate response to maximal dose of oral furosemide (>2.5 mg/kg/day) - or
  * requiring other methods of treatment [i.e. PUF or hemodialysis], based on persistence of high venous congestion (detected with central venous pressure measurement: >8 mm Hg or dilated inferior cava vein, without respiratory change, measured with focused abdominal echography, and coupled with body weight increase of 1 kg or more in the last 24 hrs.

SECONDARY OUTCOMES:
6 min Walking distance | At 3, 6 and 7 months from randomization
  Change from the baseline
Quality of life tested with Kansas City Cardiomyopathy Questionnaire (KCCQ) | At 3, 6 and 7 months from randomization
  Change from the baseline
Number of patients with decrease of NT pro-BNP (N-terminal pro brain natriuretic peptide) | At 3, 6 and 7 months from randomization
  The number of patients with a decrease in NT pro-BNP level of ≥25% from baseline
Worsening of renal function | Up to 7 months from randomization
  Estimated Glomerular Filtration Rate (eGFR) ≤20 ml/min
Cumulative daily dosage of loop diuretic | Up to 7 months from randomization
  Change over the 6 months of study treatment,
Use of hospital resources | Up to 7 months from randomization
  The number of days spent in-hospital because of HF exacerbation during the 6 months of study treatment
New York Heart Association (NYHA) class | At 3, 6 and 7 months from randomization and during long-term FUs
  Change from baseline
Number of patients requiring hospitalization | Up to 7 months from randomization
  Hospitalization for infusional therapy with loop diuretic
Number of patients increasing of ≥50% the initial daily dose of loop diuretic | Up to 7 months from randomization
  Change from baseline
Adverse Events | through study completion, an average of 1 year
  Information about all adverse events, whether volunteered by the patient, discovered by investigator questioning, or detected through physical examination, laboratory or instrumental test, will be collected, recorded and followed as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Gronda, MD, Study Director — Policlinico Milano - on behalf of Cardio Renal and Metabolism Working Group of the ANMCO
Locations (3):
- Italy (3):
  - Ospedale Ss. Annunziata, Chieti
  - ASST FBF Sacco, Milan
  - Ospedale Monaldi, Napoli

IPD SHARING:
Plan to Share IPD: No